CLINICAL TRIAL: NCT01584336
Title: Prospective Multi-center Study of Laparoscopy-assisted Total Gastrectomy for Clinical Stage I Gastric Cancer (KLASS-03)
Brief Title: Laparoscopy-assisted Total Gastrectomy for Clinical Stage I Gastric Cancer (KLASS-03)
Acronym: KLASS-03
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Gyu-Seok Cho, Soonchunhyang University Bucheon Hospital, Soonchunhyang University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KLASS-03
Record Dates: First submitted 2012-04-22; First posted 2012-04-24 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2014-02

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer, laparoscopy-assisted total gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LATG group (Experimental): It means the patients who will be enrolled in our study.
  Interventions: Procedure: LATG

INTERVENTIONS:
Procedure: LATG — 1. After laparoscopic observation, the surgeon must check the possibility of laparoscopic surgery (without the serosal invasion of cancer or peritoneal metastasis or lymph node metastasis to splenic hilum). If the gastric cancer with serosal invasion or grossly lymph node metastasis to splenic hilum, operator must convert the operation method to open gastrectomy
  2. The operator undergoes the laparoscopic total gastrectomy with lymph node dissection(including the status of lymph nodes - No #1,2,3,4sa,4sb,4d,5,6,7,8a,9,11p and 11d, and/or 12a).
  3. The operator can choose any reconstruction method of esophagojejunostomy according to surgeon's preference.
  4. After then, the operator performs the jejunojejunostomy.
  Other Names: Laparoscopy-assisted total gastrectomy (LATG)

SUMMARY:
The purpose of this study is to evaluate the safety and feasibility of laparoscopy-assisted total gastrectomy for early upper gastric cancer compared with open total gastrectomy. This study will performed via prospective, multicenter design.

DETAILED DESCRIPTION:
Gastric cancer remains one of the most common neoplasms in Asia and some western countries, although the incidence is decreasing worldwide. Recently,as the rate of detection of early gastric cancer has increased and surgical techniques have been developed, laparoscopic procedures have been introduced and tried for the treatment of early-stage gastric cancer.

Already the prospective, randomized trials for safety and oncologic outcomes of laparoscopy-assisted distal gastrectomy for gastric cancer had been tried, but the large-scaled, prospective study for laparoscopy-assisted total gastrectomy (LATG) is seldom.

One reason for the low popularity is that LATG requires the dissection of lymph nodes at the splenic hilum or along the short gastric arteries and the other reason is that the reconstruction after total gastrectomy is also more complicated. The third reason is that the chance for total gastrectomy is less frequent than distal gastrectomy because of the low incidence of upper gastric cancer.

This KLASS-03 trial is a prospective, multicenter trial for LATG for early upper gastric cancer. The primary purpose of this study is to evaluate the incidence of postoperative morbidity and mortality and the second purpose is to evaluate the surgical outcomes after several methods of reconstruction in laparoscopic total gastrectomy and the postoperative course of LATG patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically diagnosed as gastric adenocarcinoma under preoperative endoscopic biopsy
* range of age ; over 20 years to under 80 years
* preoperative stage : cT1N0M0, cT1N1M0, cT2N0M0 (7th UICC)
* The patient who is needed the total gastrectomy because the upper margin of cancer is located between upper 1cm and lower 5cm to esophagogastric junction
* the gastric cancer which is not included the indication of the endoscopic mucosal dissection
* ECOG (Eastern Cooperative Oncology Group) performance status; 0 and 1
* ASA (American Society of Anesthesiology) score ; 1, 2, 3
* Written informed consent

Exclusion Criteria:

* The patient who shows distant metastasis under preoperative examination
* The patient with medical history for upper abdominal surgery with open method in the past
* The patient with medical history for distal gastrectomy due to benign or malignant gastric disease in the past(remnant stomach cancer)
* The patient with double cancer synchronous or metachronous within 5 years
* Enlarged lymph nodes of the splenic hilum in the preoperative evaluation
* The patient who has been enrolled other clinical study within 6 months
* Vulnerable patients who lacks mental capacity and are pregnant or planning a pregnancy

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-02 (Actual); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
The incidence of postoperative morbidity and mortality | 1 month
  The primary purpose of this study is that the incidence of morbidity and mortality after LATG. We will access the postoperative morbidity including as follows: wound complication, intra-abdominal fluid collection or abscess, intra-abdominal bleeding, intraluminal bleeding, intestinal obstruction, ileus, anastomotic stenosis, anastomotic leakage, fistula, pancreatitis, pulmonary complication, urinary complication, renal complication, hepatic complication, cardiac complication, endocrine complication, and stasis.
  Also we will evaluate the incidence of postoperative mortality after LATG.

SECONDARY OUTCOMES:
the surgical outcomes according to the method of reconstruction | 1 month
  We will evaluate the difference of surgical outcomes (duration of anastomosis, failure rate of anastomosis, etc) and postoperative morbidity (anastomotic leakage, stenosis, bleeding, etc) according to the methods of reconstruction after gastrectomy. The methods of reconstruction after gastrectomy will be depend to the each operator's decision.

CONTACTS AND LOCATIONS:
Overall Officials: Gyu-Seok Cho, M.D., Ph.D., Principal Investigator — Soonchunhyang University Hospital
Locations (7):
- South Korea (7):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Keimyung University Dongsan Medical Center, Daegu
  - Kyungpook National University medical Center, Daegu
  - Incheon St, Mary's Hostpial, The Catholic University of Korea, Incheon
  - Seoul National University Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul

REFERENCES:
- [Background] Kim SG, Lee YJ, Ha WS, Jung EJ, Ju YT, Jeong CY, Hong SC, Choi SK, Park ST, Bae K. LATG with extracorporeal esophagojejunostomy: is this minimal invasive surgery for gastric cancer? J Laparoendosc Adv Surg Tech A. 2008 Aug;18(4):572-8. doi: 10.1089/lap.2007.0106. PMID 18721007
- [Background] Kunisaki C, Makino H, Oshima T, Fujii S, Kimura J, Takagawa R, Kosaka T, Akiyama H, Morita S, Endo I. Application of the transorally inserted anvil (OrVil) after laparoscopy-assisted total gastrectomy. Surg Endosc. 2011 Apr;25(4):1300-5. doi: 10.1007/s00464-010-1367-5. Epub 2010 Oct 17. PMID 20953884
- [Background] Nunobe S, Hiki N, Tanimura S, Kubota T, Kumagai K, Sano T, Yamaguchi T. Three-step esophagojejunal anastomosis with atraumatic anvil insertion technique after laparoscopic total gastrectomy. J Gastrointest Surg. 2011 Sep;15(9):1520-5. doi: 10.1007/s11605-011-1489-7. Epub 2011 May 10. PMID 21557017
- [Background] Okabe H, Obama K, Tanaka E, Nomura A, Kawamura J, Nagayama S, Itami A, Watanabe G, Kanaya S, Sakai Y. Intracorporeal esophagojejunal anastomosis after laparoscopic total gastrectomy for patients with gastric cancer. Surg Endosc. 2009 Sep;23(9):2167-71. doi: 10.1007/s00464-008-9987-8. Epub 2008 Jun 14. PMID 18553203
- [Result] Kim MG, Kim BS, Kim TH, Kim KC, Yook JH, Kim BS. The effects of laparoscopic assisted total gastrectomy on surgical outcomes in the treatment of gastric cancer. J Korean Surg Soc. 2011 Apr;80(4):245-50. doi: 10.4174/jkss.2011.80.4.245. Epub 2011 Apr 12. PMID 22066043
- [Result] Kanagale P, Lohray BB, Misra A, Davadra P, Kini R. Formulation and optimization of porous osmotic pump-based controlled release system of oxybutynin. AAPS PharmSciTech. 2007 Jul 13;8(3):E53. doi: 10.1208/pt0803053. PMID 17915803
- [Result] Mochiki E, Toyomasu Y, Ogata K, Andoh H, Ohno T, Aihara R, Asao T, Kuwano H. Laparoscopically assisted total gastrectomy with lymph node dissection for upper and middle gastric cancer. Surg Endosc. 2008 Sep;22(9):1997-2002. doi: 10.1007/s00464-008-0015-9. Epub 2008 Jul 2. PMID 18594925
- [Result] Kawamura H, Yokota R, Homma S, Kondo Y. Comparison of invasiveness between laparoscopy-assisted total gastrectomy and open total gastrectomy. World J Surg. 2009 Nov;33(11):2389-95. doi: 10.1007/s00268-009-0208-y. PMID 19760315
- [Result] Tanimura S, Higashino M, Fukunaga Y, Takemura M, Tanaka Y, Fujiwara Y, Osugi H. Laparoscopic gastrectomy for gastric cancer: experience with more than 600 cases. Surg Endosc. 2008 May;22(5):1161-4. doi: 10.1007/s00464-008-9786-2. Epub 2008 Mar 6. PMID 18322744
- [Result] Lee SE, Ryu KW, Nam BH, Lee JH, Kim YW, Yu JS, Cho SJ, Lee JY, Kim CG, Choi IJ, Kook MC, Park SR, Kim MJ, Lee JS. Technical feasibility and safety of laparoscopy-assisted total gastrectomy in gastric cancer: a comparative study with laparoscopy-assisted distal gastrectomy. J Surg Oncol. 2009 Oct 1;100(5):392-5. doi: 10.1002/jso.21345. PMID 19598150